CLINICAL TRIAL: NCT00516958
Title: An Open Label, Three Arm, Pilot Study of the Safety and Clinical Efficacy of Topical Dermacyn™ Wound Care vs. Oral Levofloxacin vs. Combined Therapy for Mild Diabetic Foot Infections
Brief Title: Pilot Study of the Safety and Clinical Efficacy of Topical Dermacyn™ Wound Care to Treat Mild Diabetic Foot Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oculus Innovative Sciences, Inc. (Industry)
Responsible Party: Andres Gutierrez, M.D., Ph.D., Oculus Innovative Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OIS-005
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Foot Ulcer, Diabetic
Keywords: diabetic; ulcer; infection; topical; wound
MeSH Terms: conditions — Diabetic Foot; Ulcer; Infections; Wounds and Injuries | interventions — dermacyn; Levofloxacin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Topical Dermacyn
  Interventions: Drug: Topical Dermacyn
- 2 (Active Comparator): Topical Dermacyn and levofloxacin
  Interventions: Drug: Topical Dermacyn and Levofloxacin
- 3 (Active Comparator): Topical saline and levofloxacin
  Interventions: Drug: Topical Saline and Levofloxacin

INTERVENTIONS:
Drug: Topical Dermacyn — Topical Dermacyn once a day for 10 Days
  Other Names: Dermacyn™ Wound Care
  Arms: 1
Drug: Topical Dermacyn and Levofloxacin — Topical Dermacyn once a day and levofloxacin 750 mg PO per day; both for 10 days
  Other Names: Dermacyn™ Wound Care; Levaquin®
  Arms: 2
Drug: Topical Saline and Levofloxacin — Topical saline once a day and levofloxacin 750 mg PO daily, both for 10 days
  Other Names: Saline Solution; Levoquin®
  Arms: 3

SUMMARY:
To compare the rates of clinical success of Topical Dermacyn™ vs. Oral Levofloxacin vs. Combined therapy, in subjects with mild diabetic foot infections in non-ischemic ulcers.

ELIGIBILITY:
Inclusion Criteria:

* A patient must meet all of the following inclusion criteria to be enrolled in the study:

  1. Males and females > 18 years of age with diabetes mellitus (type 1 or type 2, controlled).
  2. Presence of infected, non-ischemic diabetic foot ulcer that involves skin and deeper soft tissue as stratified by IDSA guidelines and the UTC / 1B.
  3. Foot infections that are anticipated to be cured in 10 days of oral antibiotic therapy.
  4. Foot ulcers located in the plantar, dorsal or malleolar areas.
  5. Ulcers 1- 9 cm2 in size.
  6. An accessible infection site for culture.
  7. ABI by Doppler ≥ 0.8 or TcPO2 ≥ 30 mmHg.
  8. Palpable pulse on the study foot (either dorsalis or posterior tibial artery).
  9. Willing and able to give informed consent.
  10. Willing to comply with the requirements for participation in the study.

Exclusion Criteria:

Patients are excluded if they meet any of the following criteria at the time of randomization:

1. Previous antibiotic treatment received for more than 24 hours within 72 hours of study.
2. Necrotizing fasciitis, deep abscesses in the soft tissue, sinus tracts, gas gangrene, or infected burns.
3. Superinfected eczema or other chronic inflammatory skin conditions (i.e., atopic dermatitis).
4. The patient´s ulcer is located on the stump of an amputated extremity.
5. The patient's ulcer is due to a non-diabetic etiology.
6. Infections complicated by the presence of prosthetic materials.
7. Osteomyelitis
8. Females of childbearing potential who are unable to take adequate contraceptive precautions or are breastfeeding.
9. Known to have liver disease, with total bilirubin > 5 times the Upper Limit of Normal (ULN); known to have neutropenia (absolute neutrophil count <500 cells/mm3).
10. Hypersensitivity to chlorine or quinolones.
11. Need for any additional concomitant systemic antibacterial agent other than the study drug(s).
12. Concomitant glucocorticoid doses (> 5mg prednisone a day or equivalent).
13. Adjuvant therapy with hyperbaric oxygen or topical formulations containing growth factors, antimicrobials or enzymatic debriders.
14. A history of diseases of immune function (HIV, chronic granulomatous disease).
15. Any medical condition that, in the investigator´s opinion, will require dose modification of Levofloxacin to less than 750 mg a day.
16. Has received an investigational agent ≤1 month prior to the baseline evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To compare the rates of clinical success (cure + improvement) of Topical Dermacyn™ vs. Oral Levofloxacin vs. Combined therapy, in patients with mild diabetic foot infections in non ischemic ulcers | Visit 3 (Day 10); Visit 4 (Day 24)

SECONDARY OUTCOMES:
To compare the treatment groups with respect to microbiological outcome. Incidence of adverse events and other safety outcomes | Visit 2 (Day 3); Visit 3 (Day 10)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Gutierrez, M.D., Ph.D., Study Director — Oculus Innovative Sciences
Locations (16):
- United States (16):
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - San Diego, California
  - Santa Rosa, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Spring Hill, Florida
  - Evansville, Indiana
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Harrisburgh, Pennsylvania
  - Hazleton, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah

REFERENCES:
- [Background] Goretti C, Mazzurco S, Nobili LA, Macchiarini S, Tedeschi A, Palumbo F, Scatena A, Rizzo L, Piaggesi A. Clinical outcomes of wide postsurgical lesions in the infected diabetic foot managed with 2 different local treatment regimes compared using a quasi-experimental study design: a preliminary communication. Int J Low Extrem Wounds. 2007 Mar;6(1):22-7. doi: 10.1177/1534734606298543. PMID 17344198
- [Background] Landa-Solis C, Gonzalez-Espinosa D, Guzman-Soriano B, Snyder M, Reyes-Teran G, Torres K, Gutierrez AA. Microcyn: a novel super-oxidized water with neutral pH and disinfectant activity. J Hosp Infect. 2005 Dec;61(4):291-9. doi: 10.1016/j.jhin.2005.04.021. Epub 2005 Oct 19. PMID 16242210
- [Background] Duc Ql, Breetveld M, Middelkoop E, Scheper RJ, Ulrich MM, Gibbs S. A cytotoxic analysis of antiseptic medication on skin substitutes and autograft. Br J Dermatol. 2007 Jul;157(1):33-40. doi: 10.1111/j.1365-2133.2007.07990.x. Epub 2007 Jun 6. PMID 17553033
- [Background] Medina-Tamayo J, Sanchez-Miranda E, Balleza-Tapia H, Ambriz X, Cid ME, Gonzalez-Espinosa D, Gutierrez AA, Gonzalez-Espinosa C. Super-oxidized solution inhibits IgE-antigen-induced degranulation and cytokine release in mast cells. Int Immunopharmacol. 2007 Aug;7(8):1013-24. doi: 10.1016/j.intimp.2007.03.005. Epub 2007 Apr 16. PMID 17570318
- [Background] Zahumensky E. [Infections and diabetic foot syndrome in field practice]. Vnitr Lek. 2006 May;52(5):411-6. Czech. PMID 16771079